CLINICAL TRIAL: NCT06973408
Title: Switching to a Healthy and Sustainable Diet for Planetary and Human Health
Brief Title: The SWITCH Dietary and Behavioural Intervention Study
Acronym: SWITCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Göteborg University (Other); Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SWITCH
Record Dates: First submitted 2025-03-20; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Dietary Behaviour; Dietary Intakes; Dietary Intervention; Metabolic Diseases; Blood Lipid Profiles; Blood Glucose Metabolism; Diet, Healthy
Keywords: Cardiometabolic health; Lifestyle intervention; Dietary adherence; Sustainable diet; Nordic diet; Metabolic risk factors; Randomized controlled trial; nevironmental impact of diet
MeSH Terms: conditions — Metabolic Diseases | interventions — Behavior Therapy; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Optimized lifestyle intervention group (Experimental): Receiving dietary advice, behavioral support, and provision of key foods.
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Food support; Behavioral: Dietary Advice
- Behavioral support intervention group (Active Comparator): Receiving dietary advice and behavioral support
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Dietary Advice
- Control group (Other): Receiving dietary advice according to the SWITCH diet.
  Interventions: Behavioral: Dietary Advice

INTERVENTIONS:
Behavioral: Behavioral Treatment — Behavioral support is designed to help participants adhere to the dietary recommendations through personalized coaching and motivational strategies. Participants engage in weekly or bi-weekly coaching sessions, either online or in person, where they receive guidance on overcoming challenges and maintaining dietary changes. The coaching incorporates evidence-based behavior change techniques, such as goal setting, self-monitoring, feedback on performance, problem-solving, and stimulus control. To further support behavior change, participants receive practical tools, including visual aids, educational videos, and structured meal planning resources. The overall goal of behavioral support is to encourage sustainable dietary habits by providing continuous encouragement and individualized strategies.
  Other Names: Behavioural support
  Arms: Behavioral support intervention group; Optimized lifestyle intervention group
Behavioral: Food support — Food support, which is provided exclusively to participants in the Optimized Lifestyle Intervention Group, ensures that they have access to key foods required to meet dietary targets. These foods include whole grains such as whole grain bread, oats, and pasta; vegetables in both fresh and frozen forms; fruits and berries, including apples, pears, and frozen berries; legumes such as lentils, beans, and chickpeas; and seafood, including fatty fish, lean fish, and mussels. To facilitate adherence, participants also receive recipes and meal plans that incorporate these foods. Some fresh food items are made available at supermarkets near participants' residences to improve accessibility and convenience. Food support aims to reduce barriers to dietary change by ensuring that participants have the necessary ingredients to follow the SWITCH diet effectively.
  Arms: Optimized lifestyle intervention group
Behavioral: Dietary Advice — Dietary advice consists of a simple document outlining the SWITCH diet, which is based on European and Nordic dietary guidelines. Participants receive this information in written form without any additional guidance, counseling, or support. The SWITCH diet emphasizes increased consumption of whole grains, vegetables, fruits, legumes, and seafood while limiting processed foods, added sugars, and excessive salt.

SUMMARY:
The overall objective of this study is to evaluate the effectiveness of an optimized lifestyle intervention based on dietary advice, behavioral support, and provision of key foods compared to dietary advice with behavioral support or dietary advice alone. The intervention aims to improve nutritional status, metabolic risk factors, and planetary sustainability.

A total of 300 participants (150 men and 150 women) who meet all inclusion criteria and none of the exclusion criteria will be recruited. The study will be conducted at the Centre for Lifestyle Intervention at Östra Hospital in Gothenburg, led by researchers from Chalmers University of Technology, University of Gothenburg, and Sahlgrenska University Hospital. Participants will be recruited from two different socioeconomic areas in Gothenburg to examine how dietary interventions function in diverse population groups.

The study follows a twelve-week randomized, controlled, parallel intervention design. Participants will be randomized into three groups, each with 100 individuals:

Optimized lifestyle intervention group - receiving dietary advice, behavioral support, and provision of key foods.

Behavioral support intervention group - receiving dietary advice and behavioral support.

Control group - receiving dietary advice according to the SWITCH diet. The SWITCH diet, developed within the EU project SWITCH, is designed to align with European dietary guidelines and promote sustainable and healthy eating habits. It emphasizes whole grains, vegetables, fruits, legumes, and sustainable seafood while limiting processed foods, added sugars, and salt.

Throughout the study, participants will undergo clinical assessments at baseline, midpoint (week 7), and endpoint (week 13). Key measurements include anthropometric data, blood pressure, blood glucose, blood lipids, and inflammatory markers. Dietary intake and sustainability aspects of food consumption will also be evaluated. Participants in the intervention groups will receive personalized coaching and access to practical resources, such as meal plans, recipes, and visual educational materials.

The primary outcome of the study is the difference in cardiometabolic risk factors (e.g., blood lipids, blood pressure, glucose, insulin resistance markers) between the intervention groups. Secondary outcomes include changes in dietary intake, nutritional status markers, inflammatory markers, and sustainability measures (e.g., CO₂ emissions, land use, biodiversity impact). Additionally, exploratory analyses will investigate associations between diet, lifestyle changes, gut microbiota, and metabolic responses.

This study aims to generate valuable insights into the effectiveness of different dietary intervention strategies in real-life Nordic conditions. The results will contribute to the development of evidence-based recommendations for sustainable and health-promoting dietary patterns.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Body mass index 25-35 kg/m2
* Stable dietary patterns at the entry to the study (no specific dieting the last 4 weeks).
* Willingness to adhere to advised diet pattern and to consume provided key foods.
* Medications stable for the previous 14 days of relevant medicines
* Access to a -18⁰ C freezer to store key foods at home.
* Signed informed consent

Exclusion Criteria:

* Currently having an infection or other relevant illness.
* Cardiovascular events (myocardial infarction or stroke) during the previous 6 months. To be included, the disease needs to be stable.
* Diagnosis of diabetes (any type).
* Blood Pressure (BP): ≥185/105 mmHg.
* Serum Cholesterol (S-Chol): ≥8 mmol/L.
* Blood Glucose (B-Glucose): fasting value >7 mmol/L.
* Currently on GLP-1 receptor agonists.
* History of stomach or gastrointestinal diagnoses (inflammatory bowel disease, Crohn's disease, hepatitis, malabsorption, celiac disease etc.).
* IBS- if severe and recent (<0.5year)?
* Previous colostomy, bowel resection, bariatric surgery or other major gastrointestinal surgery.
* Renal or liver failure (creatinine <1.7 mg/dl and alanine aminotransferase/ aspartate aminotransferase > 2 times than normal values (ASAT, ALAT), respectively).
* Anemia or Hemoglobin (Hb): <100 g/L
* Blood donation (or participation in a clinical study with blood sampling) within 30 days prior to inclusion
* Currently on a specific diet.
* A diet incompatible with protocol diets such as strict vegan/vegetarian.
* Food allergies or intolerances to food items included in the intervention.
* High level of regular physical activity at baseline - scale 4 on SG-PALS.
* History of drug or alcohol abuse.
* Not able to understand written or spoken Swedish.
* Any other reason for lack of suitability for participation in the trial, as judged by the principal investor and/ or the clinical investigator.
* Pregnant or lactating or planning to become pregnant during the study period.
* Involved in another potentially interfering research study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
LDL cholesterol | After 6 and 12 weeks of intervention
  Changes in fasting LDL cholesterol
HDL cholesterol | After 6 and 12 weeks of intervention
  Changes in fasting HDL cholesterol
non-HDL cholesterol | After 6 and 12 weeks of intervention
  Changes in fasting nonHDL cholesterol
Total cholesterol | After 6 and 12 weeks of intervention
  Changes in fasting total cholesterol
Triglyceride | After 6 and 12 weeks of intervention
  Changes in fasting triglycerides
Blood pressure | After 6 and 12 weeks of intervention
  Change in systolic and/or diastolic blood pressure
Blood glucose | After 6 and 12 weeks of intervention
  Changes in fasting blood glucose levels
Insulin | After 6 and 12 weeks of intervention
  Changes in c-peptid in fasting samples

SECONDARY OUTCOMES:
Intake of key food groups and key nutrients | After 6 and 12 weeks of intervention
  Intake of eg. whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids.
Nutritional status markers | After 6 and 12 weeks of intervention
  Eg. fatty acids, vitamin D, iron, selenium, iodine, zink, folate and B12
Planetary sustainability measurements | After 6 and 12 weeks of intervention
  Carbon footprint, cropland use, new input of N and phosphorus (P), blue water use, pesticide use, biodiversity impact, land use and ammonia emissions
Inflammatory markers | After 6 and 12 weeks of intervention
  IL-6 and CRP

OTHER OUTCOMES:
Correlation between dietary changes and gut microbiota | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and gut microbiota
Correlation between dietary changes and plasma- and urinary metabolomes | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and plasma and urinary metabolomes
Correlation between lifestyle changes and plasma- and urinary metabolomes | After 6 and 12 weeks of intervention
  Exploratory associations between lifestyle changes and plasma- and urinary metabolomes
Correlation between lifestyle changes and gut microbiota | After 6 and 12 weeks of intervention
  Exploratory associations between lifestyle changes and gut microbiota
Correlation between changes in dietary intakes and HDL | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and HDL
Correlation between changes in dietary intakes and non-HDL | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and non-HDL
Correlation between changes in dietary intakes and total cholesterol | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and total cholesterol
Correlation between changes in dietary intakes and triglycerides | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and triglycerides
Correlation between changes in dietary intakes and blood pressure | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and systolic and diastolic blood pressure
Correlation between changes in dietary intakes and blood glucose | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and and blood glucose
Correlation between changes in dietary intakes and blood glucose | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and blood glucose
Correlation between changes in dietary intakes and insulin | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and insulin
Correlations between changes in dietary intakes and behavioral outcomes | After 6 and 12 weeks of intervention
  Correlation between changes in dietary intakes (whole grains, marine foods, legumes, fruits and vegetables, red and processed meats, dairy foods, sugar, starch, protein, dietary fibre, micronutrients and minerals, fatty acids) and behavioral outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Lifestyle Interventions, Sahlgrenska University Hospital, Östra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided